CLINICAL TRIAL: NCT06280638
Title: Computed Tomography Coronary Physiology-derived Virtual Stenting Guided Revascularization Strategy in Patients With Coronary Artery Disease
Brief Title: CT-derived Virtual Stenting Optimize Coronary Revascularization (CT-COMPASS)
Acronym: CT-COMPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Kefei Dou, MD, Kefei Dou, MD, Professor, China National Center for Cardiovascular Diseases, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-2095
Record Dates: First submitted 2024-02-11; First posted 2024-02-28 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Percutaneous Coronary Intervention; Coronary Physiology; Computed Tomography
Keywords: Percutaneous Coronary Intervention; Coronary Physiology; Computed Tomography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual stenting-guided incremental optimization strategy (VIOS) (Experimental): Virtual Stenting analysis is conducted based on pre-PCI CCTA angiograms by "Imaging-Heart Team" to determine simulated optimal treatment strategy according VIOS protocol. If the patient is assigned to the VIOS, the result of virtual stenting and recommended treatment strategy will be disclosed to the operator. The operator will then follow the recommended strategy to attempt to obtain the target optimal post-PCI FFR result. Blinded FFR must be obtained after PCI.
  Interventions: Other: Virtual stent-guided incremental optimization strategy (VIOS)
- Standard angiographic strategy (Sham Comparator): Virtual Stenting analysis is conducted based on pre-PCI CCTA angiograms by "Imaging-Heart Team" to determine simulated optimal treatment strategy according VIOS protocol. If the patient is assigned to the standard angiographic strategy, the result of virtual stenting and recommended treatment strategy will be blinded to the operator. The operator will then perform PCI based on international guidelines, local protocols and practice. Blinded FFR must be obtained after PCI.
  Interventions: Other: Standard angiographic strategy

INTERVENTIONS:
Other: Virtual stent-guided incremental optimization strategy (VIOS) — PCI is performed according to strategy recommended by "Imaging-Heart Team" based on VIOS protocol.
  Other Names: VIOS-based PCI
  Arms: Virtual stenting-guided incremental optimization strategy (VIOS)
Other: Standard angiographic strategy — PCI is performed based on international guidelines, local protocols and practice.
  Other Names: angio-based PCI
  Arms: Standard angiographic strategy

SUMMARY:
A considerable number of patients presented with anatomically successful PCI results still suffer from functionally unresolved ischemia, which might be the cause for over one-fourth of patients experiencing recurrent angina at 1 year or adverse events at 2 years. Currently, the post-PCI physiology measurement is one of the effective metrics to quantify residual ischemia, and a suboptimal post-PCI result is strongly associated with worse outcomes. However, PCI optimization based on post-PCI physiology is, to certain extent, a provisional rescue action for a suboptimal index procedure, which may not be fully correctable "after the fact" given selected stents, site of deployment and procedural technique.

Computed tomography (CT) coronary physiology-derived virtual stenting (CT-VS) based on pre-PCI CCTA angiograms is an augmented reality (AR) approach that simulates the post-stenting physiology assuming that the specified segment of the treated vessel is successfully dilated by implanting virtual stents. Previous studies have demonstrated the feasibility of optimizing PCI with CT-VS, with high consistency between pre-PCI simulated physiology result by CT-VS and actual post-PCI physiology results. Therefore, the application of CT-VS would help physicians to develop the best strategies while planning the procedure.

However, there is a lack of knowledge regarding the efficacy of this novel physiological index that is available pre-PCI in achieving final post-PCI optimal physiological result. The Trials of "Computed Tomography Coronary Physiology-derived Virtual Stenting Guided Revascularization Strategy in Patients with Coronary Artery Disease (CT-COMPASS)" was designed to assess the efficacy of a CT-VS vs. standard angiographic guidance in achieving post-PCI optimal physiological result (post-PCI FFR≥0.90).

DETAILED DESCRIPTION:
Coronary physiology-guided percutaneous coronary intervention (PCI) improves long-term prognosis in large clinical studies, and wire-based physiological assessments (e.g. fractional flow reserve [FFR], instantaneous wave-free ratio [iFR]) are recommended by international guidelines. Although prognosis of patients undergoing PCI has improved in recent decades with the continuous refinement of equipment, tools and techniques, a considerable number of patients presented with anatomically successful PCI results still suffer from functionally unresolved ischemia, which might be the cause for over one-fourth of patients experiencing recurrent angina or adverse events after angiographically successful PCI. Therefore, it is of great clinical importance to achieve complete resolution of ischemia and optimal functional results during the index procedure.

Currently, the post-PCI physiology measurement is one of the effective metrics to quantify residual ischemia, and a suboptimal post-PCI result is strongly associated with worse outcomes. However, PCI optimization based on post-PCI physiology is, to certain extent, a provisional rescue action for a suboptimal index procedure, which may not be fully correctable "after the fact" given selected stents, site of deployment and procedural technique. The resent TARGET-FFR trial demonstrated that post-PCI physiology-guided incremental optimization strategy (PIOS) failed to significantly improve the final physiological results compared to standard angiographic guidance. Therefore, it would be of significant interest if a preprocedural measurement would be able to anticipate to what extent the functional ischemia could be resolved. If residual ischemia estimated from the computation of post-PCI physiology appears to be present, this would help physicians to develop the best strategies while planning the procedure.

The Computed tomography (CT)-derived FFR (CT-FFR) is a novel non-invasive CCTA-based physiological index that has been validated to have good diagnostic accuracy in identifying physiologically significant coronary stenoses compared with FFR as the reference. The CT coronary physiology-derived virtual stenting (CT-VS) based on pre-PCI CCTA angiograms, is an augmented reality (AR) approach that simulates the post-stenting physiology assuming that the specified segment of the treated vessel is successfully dilated by implanting virtual stents. Previous studies have demonstrated the feasibility of optimizing PCI with CT-VS, with high consistency between pre-PCI simulated physiology result by CT-VS and actual post-PCI physiology results. Therefore, the application of CT-VS would help physicians to develop the best strategies while planning the procedure.

However, there is a lack of knowledge regarding the efficacy of this novel physiological index that is available pre-PCI in achieving final post-PCI optimal physiological result. The Trials of "Computed Tomography Coronary Physiology-derived Virtual Stenting Guided Revascularization Strategy in Patients with Coronary Artery Disease (CT-COMPASS)" was designed to assess the efficacy of a CT-VS vs. standard angiographic guidance in achieving post-PCI optimal physiological result (post-PCI FFR≥0.90).

Virtual stenting-guided incremental optimization strategy (VIOS) Protocol: virtual Stenting analysis is conducted based on pre-PCI CCTA angiograms by "Imaging-Heart Team" to determine simulated optimal treatment strategy according VIOS protocol. The details of VIOS protocol are as follows: 1) virtual stent with adequate stent parameters is initially implanted to treat lesion with maximal CT-FFR drop (ΔCT-FFR); 2) if the simulated post-PCI CT-FFR is ≥0.90, no further intervention will be performed, and the simulated optimal treatment strategy is determined. If simulated post-PCI CT-FFR is <0.90, the "Imaging-Heart Team" would then have the following options: a) if there is a CT-FFR drop ≥0.05 across the virtual stented segment(s), the parameters of virtual stent(s) would be optimized (i.e., number of stents, stent diameter, and stent length); b) if there is a CT-FFR drop ≥0.05 across a relatively focal (<20mm) unstented segment (without virtual stenting) which is suitable for further stenting then a further virtual stent would be implanted; c) simulated post-PCI CT-FFR remains <0.90 after steps a and/or b: if either of the above criteria remain, option of further optimization of virtual stent parameters or one more additional virtual stent. Following this, the result will be accepted. d) if the simulated CT-FFR gradient is interpreted to reflect diffuse atherosclerosis with no focal CT-FFR drop, the result is accepted.

ELIGIBILITY:
Inclusion Criteria

General Inclusion Criteria

1. Age ≥ 18 years.
2. Able to understand the trial design and provide written informed consent.
3. Patients with a coronary CTA performed within 30 days.

CCTA Inclusion Criteria

1. The CCTA angiograms amenable to CT-FFR measurement.
2. At least 1 lesion of 50%-90% diameter stenosis in a coronary artery with ≥2.0mm reference vessel diameter by visual assessment.
3. And this target vessel is of physiological ischemia as assessed by CT-FFR.

Angiographic Inclusion Criteria

1. The interrogated vessel is indicated for intervention assessed by operator based on indications other than CT-FFR.

Exclusion Criteria

General Exclusion Criteria

1. Cardiogenic shock or severe heart failure (NYHA ≥III or LVEF<30%).
2. Severely impaired renal function: creatinine >150μmol/L or Cockcroft-Gault calculated GFR <45 ml/kg/1.73 m2 (calculated with Cockcroft-Gault formula).
3. Allergy to iodine-containing contrast agents which cannot be adequately premedicated.

CCTA Exclusion Criteria

1. The CCTA angiograms deems not amenable to CT-FFR measurement.
2. Patients with only 1 coronary artery lesion with DS >90% with TIMI flow <3.
3. An interrogated vessel presented with a CTO lesion.
4. All coronary arteries were not physiologically ischemic.
5. Coronary lesions favor CABG treatment.

Angiographic Exclusion Criteria

1. The interrogated vessel with only 1 coronary artery lesion with DS >90% with TIMI flow <3.
2. Coronary lesions favor CABG treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with a final post-PCI FFR result ≥0.90 | 1 days
  The proportion of patients with a final post-PCI FFR result ≥0.90 will be compared between the randomised groups

SECONDARY OUTCOMES:
The proportion of patients with final post-PCI FFR ≤0.80 | 1 days
  The proportion of patients with a final post-PCI FFR result ≤0.80 will be compared between the randomised groups
The rate of target vessel failure (TVF) and its component features at 6 months. | 6 months
  Component features of TVF include cardiac death, target vessel myocardial infarction, and target vessel revascularisation.
The rate of target vessel failure (TVF) and its component features at 1 year. | 1 year
  Component features of TVF include cardiac death, target vessel myocardial infarction, and target vessel revascularisation.
Change from baseline in self-reported Health-related quality of life evaluation at 6 months. | 6 months
  Patients will complete the European Quality of Life-5 Dimensions (EQ-5D) questionnaire at baseline pre-procedure and again at 6 months post PCI
Change from baseline in self-reported Health-related quality of life evaluation at 1 year. | 1 year
  Patients will complete the European Quality of Life-5 Dimensions (EQ-5D) questionnaire at baseline pre-procedure and again at 1 year post PCI
Change from baseline in self-reported Angina status evaluation at 6 months. | 6 months
  Patients will complete the Seattle Angina Questionnaire (SAQ) at baseline pre-procedure and again at 6 months post PCI
Change from baseline in self-reported Angina status evaluation at 1 year. | 1 year
  Patients will complete the Seattle Angina Questionnaire (SAQ) at baseline pre-procedure and again at 1 year post PCI
Procedure Duration | 1 day
  The time required to perform the VIOS intervention procedures will be compared with those in the control group.
Fluoroscopy Dose | 1 day
  The radiation doses for the VIOS intervention procedures will be compared with those in the control group.
Contrast Material Dose | 1 day
  The contrast material doses for the VIOS intervention procedures will be compared with those in the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Kefei Dou, MD, PhD, Principal Investigator — Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Sonck J, Nagumo S, Norgaard BL, Otake H, Ko B, Zhang J, Mizukami T, Maeng M, Andreini D, Takahashi Y, Jensen JM, Ihdayhid A, Heggermont W, Barbato E, Mileva N, Munhoz D, Bartunek J, Updegrove A, Collinsworth A, Penicka M, Van Hoe L, Leipsic J, Koo BK, De Bruyne B, Collet C. Clinical Validation of a Virtual Planner for Coronary Interventions Based on Coronary CT Angiography. JACC Cardiovasc Imaging. 2022 Jul;15(7):1242-1255. doi: 10.1016/j.jcmg.2022.02.003. Epub 2022 Apr 13. PMID 35798401
- [Background] Biscaglia S, Verardi FM, Tebaldi M, Guiducci V, Caglioni S, Campana R, Scala A, Marrone A, Pompei G, Marchini F, Scancarello D, Pignatelli G, D'Amore SM, Colaiori I, Demola P, Di Serafino L, Tumscitz C, Penzo C, Erriquez A, Manfrini M, Campo G. QFR-Based Virtual PCI or Conventional Angiography to Guide PCI: The AQVA Trial. JACC Cardiovasc Interv. 2023 Apr 10;16(7):783-794. doi: 10.1016/j.jcin.2022.10.054. Epub 2023 Mar 8. PMID 36898939
- [Background] Collison D, Didagelos M, Aetesam-Ur-Rahman M, Copt S, McDade R, McCartney P, Ford TJ, McClure J, Lindsay M, Shaukat A, Rocchiccioli P, Brogan R, Watkins S, McEntegart M, Good R, Robertson K, O'Boyle P, Davie A, Khan A, Hood S, Eteiba H, Berry C, Oldroyd KG. Post-stenting fractional flow reserve vs coronary angiography for optimization of percutaneous coronary intervention (TARGET-FFR). Eur Heart J. 2021 Dec 1;42(45):4656-4668. doi: 10.1093/eurheartj/ehab449. PMID 34279606
- [Background] Zhang R, Xu B, Dou K, Guan C, Zhao Y, Wang X, Zou T, Qiao Z, Xie L, Wang H, Yuan S, Song L, Tu S, Wang Y, Wijns W. Post-PCI outcomes predicted by pre-intervention simulation of residual quantitative flow ratio using augmented reality. Int J Cardiol. 2022 Apr 1;352:33-39. doi: 10.1016/j.ijcard.2022.01.054. Epub 2022 Jan 31. PMID 35101540
- [Background] Xu B, Tu S, Song L, Jin Z, Yu B, Fu G, Zhou Y, Wang J, Chen Y, Pu J, Chen L, Qu X, Yang J, Liu X, Guo L, Shen C, Zhang Y, Zhang Q, Pan H, Fu X, Liu J, Zhao Y, Escaned J, Wang Y, Fearon WF, Dou K, Kirtane AJ, Wu Y, Serruys PW, Yang W, Wijns W, Guan C, Leon MB, Qiao S, Stone GW; FAVOR III China study group. Angiographic quantitative flow ratio-guided coronary intervention (FAVOR III China): a multicentre, randomised, sham-controlled trial. Lancet. 2021 Dec 11;398(10317):2149-2159. doi: 10.1016/S0140-6736(21)02248-0. Epub 2021 Nov 4. PMID 34742368
- [Background] Ding D, Huang J, Westra J, Cohen DJ, Chen Y, Andersen BK, Holm NR, Xu B, Tu S, Wijns W. Immediate post-procedural functional assessment of percutaneous coronary intervention: current evidence and future directions. Eur Heart J. 2021 Jul 15;42(27):2695-2707. doi: 10.1093/eurheartj/ehab186. PMID 33822922
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437